CLINICAL TRIAL: NCT00594412
Title: Validation of (1)H-Magnetic Resonance Spectroscopy for Quantification of Hepatic Triglyceride Content
Brief Title: MRI to Measure Liver Fat Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 080034; 08-I-0034
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-06-15

CONDITIONS: Fatty Liver; Hepatitis
Keywords: 1H-Magnetic Resonance Spectroscopy; Hepatic Steatosis; Liver Fat; Liver Biopsy; Liver; Hepatitis; Fatty Liver
MeSH Terms: conditions — Fatty Liver; Hepatitis

INTERVENTIONS:
Procedure: Diagnostic Radiology: 1H-MRS of the liver

SUMMARY:
This study will determine whether a magnetic resonance imaging (MRI) test of the liver can accurately measure the amount of fat in the liver compared to the results of a liver biopsy.

People 18 years of age and older who are scheduled to have or who have already had a liver biopsy as part of their medical care within 1 month of enrollment in this study may be eligible to participate.

Participants undergo an MRI. For this procedure, the subject lies still on a table that slides into a narrow metal cylinder (the MRI scanner) for 30 to 60 minutes. A special pad or tube is placed around the abdomen to improve the image of the liver obtained. Earplugs are placed in the ears to muffle loud thumping and knocking sounds that occur with the electrical switching of the magnetic field. The findings of the MRI are compared with those of the liver biopsy.

DETAILED DESCRIPTION:
Percutaneous liver biopsy remains the gold standard test to evaluate hepatic fat content, fibrosis and cirrhosis, but there is growing interest in the application of magnetic resonance imaging (MRI) techniques such as (1)H-Magnetic Resonance Spectroscopy ((1)H-MRS) as a non-invasive approach to quantify these characteristics. The ability to accurately quantify hepatic metabolites, such as intrahepatic lipid, has important implications for clinical evaluation and management of patients with liver related diseases and may obviate the need for liver biopsies in a number of clinical settings. The current proposal is designed to develop and validate hepatic (1)H-MRS capabilities at the NIH Clinical Center and to use this technique in a subsequent study to estimate the prevalence of hepatic steatosis among persons living with HIV/AIDS. In the present study we propose to complete MRI with (1)H-MRS in 70 adults who will be undergoing percutaneous liver biopsy in order to establish the ability of (1)H-MRS to accurately assess hepatic fat content compared to histopathological scoring.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18+, male or female

Planned liver biopsy or liver biopsy within the past month with pathology samples available to be read at NIH CC

EXCLUSION CRITERIA:

Known current pregnancy or pregnancy within 6 months

Contraindications to MRI

Subject is deemed unable to comply with requirements of study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-12-20; Primary Completion 2010-07-01 (Actual); Study Completion 2011-06-15 (Actual)

PRIMARY OUTCOMES:
Validate 1H-Magnetic Resonance Spectroscopy to assess hepatic steatosis

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nakao K, Nakata K, Ohtsubo N, Maeda M, Moriuchi T, Ichikawa T, Hamasaki K, Kato Y, Eguchi K, Yukawa K, Ishii N. Association between nonalcoholic fatty liver, markers of obesity, and serum leptin level in young adults. Am J Gastroenterol. 2002 Jul;97(7):1796-801. doi: 10.1111/j.1572-0241.2002.05846.x. PMID 12135038
- [Background] Banerji MA, Buckley MC, Chaiken RL, Gordon D, Lebovitz HE, Kral JG. Liver fat, serum triglycerides and visceral adipose tissue in insulin-sensitive and insulin-resistant black men with NIDDM. Int J Obes Relat Metab Disord. 1995 Dec;19(12):846-50. PMID 8963350
- [Background] Sabir N, Sermez Y, Kazil S, Zencir M. Correlation of abdominal fat accumulation and liver steatosis: importance of ultrasonographic and anthropometric measurements. Eur J Ultrasound. 2001 Dec;14(2-3):121-8. doi: 10.1016/s0929-8266(01)00153-7. PMID 11704429
- [Derived] Georgoff P, Thomasson D, Louie A, Fleischman E, Dutcher L, Mani H, Kottilil S, Morse C, Dodd L, Kleiner D, Hadigan C. Hydrogen-1 MR spectroscopy for measurement and diagnosis of hepatic steatosis. AJR Am J Roentgenol. 2012 Jul;199(1):2-7. doi: 10.2214/AJR.11.7384. PMID 22733887